CLINICAL TRIAL: NCT02239978
Title: Effect of Levodopa on Postural Motor Learning in Parkinson Disease
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: N1480-M
Record Dates: First submitted 2014-09-02; First posted 2014-09-15 (Estimated); Results first posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Posture Balance; Learning; Dopamine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — No Biospecimens will be collected or retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinsons disease: Individuals with Parkinsons disease
  Interventions: Behavioral: Postural perturbation
- Control: Age-matched healthy adults
  Interventions: Behavioral: Postural perturbation

INTERVENTIONS:
Behavioral: Postural perturbation — Participants will undergo between 50 and 100 postural perturbations (quick movements of the support surface) in multiple directions. These perturbations will be between 9 and 24cm, and between 18 and 56 cm/s depending on participant tolerance.

SUMMARY:
The primary goal of this project is to gain a better understanding of whether and how levodopa (a common anti-Parkinson disease medication) alters postural motor learning in people with Parkinson disease. A secondary goal is to assess whether motor cortical excitability, measured via Transcranial magnetic stimulation, is related to postural motor learning.

Participants with Parkinson disease will complete between 50 and 100 postural perturbations (via support surface translations), ON and OFF their dopamine replacement therapy (i.e. levodopa). Adaptation of responses to these perturbations will be tracked. Participants will also undergo transcranial magnetic stimulation to capture cortical excitability of the brain (in particular the motor cortex). Cortical excitability will be correlated to adaptation of stepping (i.e. postural motor learning) ON and OFF levodopa. Investigators will also capture postural motor learning and cortical excitability in age-matched healthy adults.

Investigators hypothesize that dopamine will have a negative effect on postural motor learning, and the cortical excitability will be correlated to postural motor learning.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 90 years of age.
* Individuals with Parkinson Disease
* Healthy adults age-matched to PD participants
* Participants with PD will be currently taking dopamine replacement (i.e. Levodopa)

Exclusion Criteria:

All subjects exclusion criteria:

* Deep brain stimulation
* Recent (within 6 months) orthopedic injuries influencing standing or balance
* Inability to stand independently

Transcranial magnetic stimulation exclusion criteria (for the subset of individuals taking part in the Transcranial Magnetic Stimulation portion of the study):

* History of epilepsy or currently taking any epileptic medication,
* History of seizures
* Family history of epilepsy or seizures

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Parkinson Disease or age-matched healthy adults in the north west United States (Oregon and Washington state).
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2016-01 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Peterson, PhD MS BS, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (3):
- United States (3):
  - Oregon Health & Science University, Portland, Oregon
  - VA Portland Health Care System, Portland, OR, Portland, Oregon
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 42 individuals were enrolled in the study (30 people with Parkinson's disease and 12 healthy older adults)
Period: Overall Study
Arm/Group | Parkinsons Disease | Control
Started | 30 | 12
Completed | 28 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parkinsons Disease | Control | Total
Number analyzed (Participants) | 30 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 14
  >=65 years | 19 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.05 (9.67) | 68.04 (6.62) | 67.16 (7.10)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 6 | 16
  Male | 20 | 6 | 26
Region of Enrollment [Number; unit: participants]
  United States | 30 | 12 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Movement of Center of Mass (COM) After Postural Perturbation
Description: Investigators will assess (via automated and custom Matlab software) the magnitude of COM movement after a postural perturbation is delivered via motion of the support surface. This will be measured throughout the intervention, as well as at follow up (24 hour later).
Time Frame: Baseline and follow up (24 hours later) both ON and OFF antiparkinson medication
Population: We were unable to collect reliable data on some of the people with PD while OFF medication, which is why there is a discrepancy between the "Parkinson's disease" and "Parkinson's disease Off Medication" arms.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Parkinson's Disease Off Medication: These are the same individuals in the "Parkinson's disease" group, but Off their levodopa
Arm/Group | Parkinsons Disease | Control | Parkinson's Disease Off Medication
Number analyzed (Participants) | 28 | 12 | 24
meters
  Start Train | 0.31 (0.11) | 0.28 (0.05) | 0.32 (0.13)
  End Train | 0.26 (0.10) | 0.23 (0.03) | 0.31 (0.12)

2. Primary Outcome: Change in Steps After Postural Perturbation
Description: Investigators will assess (via automated and custom Matlab software) the number of steps taken after a postural perturbation is delivered via motion of the support surface. This will be measured throughout the intervention, as well as at follow up (24 hour later).
Time Frame: Baseline and follow up (24 hours later) both ON and OFF antiparkinson medication
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of steps
Arm/Group | Parkinsons Disease | Control | Parkinson's Disease Off Medication
Number analyzed (Participants) | 28 | 12 | 24
Number of steps
  Start Train | 2.22 (0.9) | 2.03 (0.63) | 2.09 (0.77)
  End Train | 1.92 (1.15) | 1.15 (0.28) | 2.05 (1.12)

3. Secondary Outcome: Change in First Step Length
Description: Investigators will assess (via automated and custom Matlab software) the length of the first step after a postural perturbation is delivered via motion of the support surface. This will be measured throughout the intervention, as well as at follow up (24 hour later).
Time Frame: Baseline and follow up (24 hours later) both ON and OFF antiparkinson medication
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Parkinsons Disease | Control | Parkinson's Disease Off Medication
Number analyzed (Participants) | 28 | 12 | 24
meters
  Start of Training | 0.18 (0.06) | 0.25 (0.11) | 0.21 (0.08)
  End of Training | 0.20 (0.08) | 0.27 (0.08) | 0.21 (0.08)

4. Secondary Outcome: Cortical Excitability
Description: Investigators will assess the cortical excitability of the primary motor cortex in a subset of participants both ON and OFF levodopa. Specifically, we used transcranial magnetic stimulation to stimulate the motor cortex, where we measure muscular activity of the arm (i.e. motor evoked potentials; MEPs). The primary outcome variable noted below is the lowest stimulation setting (measured as a percentage) which results in an MEP in 5 of 10 trials.
Time Frame: TMS data was collected ON and OFF medication during one visit. This visit occurred within 3 weeks of the initial postural control assessments.
Population: As noted in our protocol, TMS was assessed in a subgroup of participants with PD. Seven of the 28 PD participants and 0 of the "control" group (healthy adults) were assessed. PD participants were assessed ON and OFF levodopa. We chose this approach because 1) this aim was exploratory in nature, and 2) MEPs of healthy adults are well characterized.
Measure: Mean (Standard Deviation); unit: % max stim output
Groups:
- Parkinson's Disease Off Medication: These are the same participants as in the Parkinson's disease group, assessed "Off" their levodopa medication
Arm/Group | Parkinsons Disease | Parkinson's Disease Off Medication
Number analyzed (Participants) | 7 | 7
% max stim output | 40.57 (8.73) | 40.71 (9.97)

ADVERSE EVENTS:
Arm/Group | Parkinsons Disease | Control
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/12
Other Adverse Events (participants affected / at risk) | 0/30 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes